CLINICAL TRIAL: NCT03142074
Title: BIOMECHANICAL AND MICROSTRUCTURAL PROPERTIES OF THE AORTIC WALL: A Pilot Study in Patients Undergoing Surgery for Ascending Aortic Aneurysms
Brief Title: Biomechanical and Microstructural Properties of Ascending Aortic Aneurysms
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59521
Record Dates: First submitted 2016-10-06; First posted 2017-05-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Aortic Aneurysms
Keywords: Improve diagnosis
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Aneurysmatic tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ascending thoracic aortic aneurysm: Biomechanical and microstructural analysis of ATAA
  ECG-gated CT
  Interventions: Other: Biomechanical and microstructural analysis of ATAA; Radiation: ECG-gated CT

INTERVENTIONS:
Other: Biomechanical and microstructural analysis of ATAA — Tissue collection; microstructural testing of tissue; mechanical testing of tissue .
Radiation: ECG-gated CT — Image analysis of ECG-gated CT.

SUMMARY:
An aortic aneurysm (thoracic or abdominal) is a permanent dilatation of the aorta caused by weakening in the arterial wall. The feared complication is aortic rupture or dissection, leading to potentially lethal aortic bleeding and associated with mortality rates up to 95%. The current diagnosis criteria do not suffice, therefore the goal of this study is the development of an improved biomechanics-based and microstructural-based diagnostic tool.

DETAILED DESCRIPTION:
An aortic aneurysm (thoracic or abdominal) is a permanent dilatation of the aorta caused by weakening in the arterial wall. The feared complication is aortic rupture or dissection, leading to potentially lethal aortic bleeding and associated with mortality rates up to 95%. Diagnosis of the aneurysm and especially its risk of rupture or dissection is highly challenging. If the aneurysm diameter and/or growth rate exceed a specific threshold (respectively 55 mm and 1 cm/year), a highly invasive and dangerous surgery is performed. However, several studies have shown no correlation between the maximum transverse diameter and the risk of rupture or dissection. Since aneurysm rupture is associated with multiple aortic tissue properties, both biomechanics-based and microstructurally-based criteria can be a promising alternative.

The overall goal of this trial is a biomechanical and microstructural analysis of aneurysms to improve the diagnostic criterion for aneurysm rupture risk. Within this goal, two scientific objectives can be distinguished. Firstly, a highly unique dataset with patient data allowing the development of an improved diagnostic tool will be created. This dataset will contain an abundance of relevant parameters such as patient characteristics, geometry, material properties and biomechanical and microstructural characteristics. The biomechanical and microstructural data will be obtained by the analysis of resected aneurysmal tissue and by dynamic imaging (4D CT). 4D CT scans are a series of ECG-gated scans that are taken at specified intervals in the cardiac circle. The second objective is to create a personalized diagnostic tool. An aneurysm rupture risk criteria based on geometry as well as biomechanical and microstructural properties is expected to be significantly more reliable than the current criteria. More specifically, a correlation between patient characteristics that can be measured non-invasively and the aneurysm rupture risk is searched for.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from thoracic aortic aneurysms (ATAA), asymptomatic or symptomatic.
* Patients with ruptured ATAA undergoing an emergency surgery.
* Signed informed consent.

Exclusion Criteria:

* Patients with ruptured ATAA due to trauma.
* The presence of any aneurysm feature that will prevent the collection of tissue samples suitable for the biomechanical and microstructural studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ATAA
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Data collection of patients suffering from thoracic aortic aneurysms | 6 years
  General information (age, gender, height, weight, BMI); medicinal usage (beta-blockers, ACE inhibitors, statins, angiotensin receptor blockers, ...); cardiovascular risk factors (smoking, hypertension, dyslipidemia, diabetes, atrial fibrillation); cardiovascular properties (tricuspid aortic valve, inherited aortopathies, abdominal aortic aneurysm, prior open heart surgery, ...)

SECONDARY OUTCOMES:
Investigation of correlation between rupture risk and mechanical and microstructural parameters | 6 years
  Mechanical properties (linear and non-linear stiffness) and histological properties (elastin fraction, collagen fraction, inflammation status, wall thickness)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Meuris, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided